CLINICAL TRIAL: NCT03886870
Title: Does Adding A Work Intervention Into An Already Existing Life Style Intervention Improve Work Ability? A Randomized Controlled Trial Study
Brief Title: Obesity, Lifestyle and Work Intervention
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Molde University College (Other)
Collaborators: Norwegian Labour and Welfare Administration (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: 2014/697 REK South-East
Record Dates: First submitted 2019-03-14; First posted 2019-03-22 (Actual); Last update posted 2019-03-22 (Actual); Status verified 2019-03

CONDITIONS: Obesity; Morbid Obesity; Sick-leave; Work Related Illnesses; Life Style
Keywords: Obesity; Work Focus; Workability; Life-style treatment
MeSH Terms: conditions — Obesity; Obesity, Morbid

STUDY DESIGN:
Intervention Model Description: The study was designed as a randomized controlled study with an exploring prospective design. The intervention lasted 12 months and each patient had three visits (baseline, 6 and 12 month) at Muritunet, each lasting 4-2-2 weeks. The participants was randomized either into a lifestyle and work intervention or into a lifestyle intervention.
  Data material gathered at each stay consisting of self-reported forms, test, journal and individual interviews. These were all collected at baseline, and at six and twelve months.
Who Masked: Participant
Masking Description: Single blind masking
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Lifestyle and work intervention (Experimental): Lifestyle intervention with work focus.
  Interventions: Behavioral: Lifestyle intervention
- Lifestyle intervention (Experimental): Lifestyle intervention without work focus.
  Interventions: Behavioral: Lifestyle and work intervention

INTERVENTIONS:
Behavioral: Lifestyle and work intervention — The intervention period lasted for a year with three institution-based stays, 4 weeks at baseline and 2 weeks at 6 and 12 months. At baseline, participants got a functional assessment and an individual adjusted rehabilitation plan. At all three stages: The intervention contains activity training with a focus on the joy of movement, strength- and cardio-training. There were lectures and cognitive therapy to promote self-care and lifestyle change. The intervention contained lectures on diet, nutrition and cooking-classes. Participants set goals at baseline and adjusting these during the progress. Exercise programs was designed to use at home. The Cognitive Information Processing model of career guidance was the mainframe for the work dimension. All participants had talks with the work consultant at baseline, 6 and 12 months. Two work lectures, "Duties and rights as employees" and "Work as medicine". When needed the work consultant contacted the employer in order to facilitate changes.
  Arms: Lifestyle intervention
Behavioral: Lifestyle intervention — The intervention period lasted for a year with three institution-based stay, 4 weeks at baseline and 2 weeks at 6 and 12 months. At baseline, participants got a functional assessment and an individual adjusted rehabilitation plan.
  At all three stages: The intervention contains activity training with focus on joy of movement, strength- and cardio-training. There was lectures and cognitive therapy to promote self-care and lifestyle change. The intervention contained lectures on diet, nutrition and cooking-classes. Participants set goals at baseline and adjusting these during the progress. They developed exercise programs designed to use at home.
  Arms: Lifestyle and work intervention

SUMMARY:
The main aim of this study was to examine whether introducing a work intervention into a traditional lifestyle rehabilitation program for persons with BMI above 30, would affect the participants' ability to work and their lifestyle change. The investigators wanted to find out how the participants experienced their health, workability and work capacity, quality of life, diet and self-efficacy before and during the intervention

DETAILED DESCRIPTION:
The background for this study was insights about obesity and sick leave. Obesity is related to lower labor force participation, increased sickness absence and reduced productivity. A Danish study from 2006 reported a yearly 1, 8 million extra days of work absence and close to 1.100 cases of disability pension related to obesity. A 2016-report from OECD show that persons with obesity between the ages 50-59 have three times as much work absence as those who do not struggle with obesity. This indicates that persons with obesity are a group where the need for work rehabilitation is important. Despite this connection, work focus has not been a part of lifestyle interventions for persons with morbid obesity until the last two years.

By introducing a work intervention into a traditional lifestyle rehabilitation program for persons with BMI over 30, the investigators wanted to examine whether this would affect the participants' ability to work and their lifestyle change. The study was designed as a randomized controlled study with an exploring prospective design. The intervention lasted 12 months and each patient had three visits (baseline, 6 and 12 months) at Muritunet, each lasting 4-2-2 weeks. The participants were randomized into two intervention, one with work intervention and one without.

Data material gathered at each stay consisting of self-reported forms, test, journal and individual interviews. These were all collected at baseline, and at six and twelve months.

ELIGIBILITY:
Inclusion Criteria:

* Participants with a Body Mass Index (BMI) > 30 with or without comorbidity

Exclusion Criteria:

* People without a capacity to consent.
* People with severe alcohol and/or drug abuse.
* People with a major mental illness.
* Being pregnant.
* People with a health condition that contraindicates physical activity.
* People with or plan to apply for disability benefits.
* People with permanently adapted work.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Actual)
Dates: Start 2014-09-03 (Actual); Primary Completion 2017-12-31 (Actual); Study Completion 2018-02-01 (Actual)

PRIMARY OUTCOMES:
Full or partial return to work. | Data collected during the interventions, baseline, 6 and 12 months.
  Mapping changes in work employability and work related factors with survey data from the ARR form (http://www.arbeidoghelse.no).

SECONDARY OUTCOMES:
Weight loss (kilograms) | Data collected during the interventions, baseline, 6 and 12 months.
  Measured changes with Tanita MC-780U Multi Frequency Segmental Body Composition Analyzer.
Return to work self-efficacy | Data collected during the interventions, baseline, 6 and 12 months.
  Mapping changes with the Return-to-work-efficacy scale (RTWSE-19). The 19-item RTWSE-19 scale is a new self-report measure intended to assess workers' beliefs of their current ability to resume normal job responsibilities following pain onset. Response range (1-10). 1 is "not sure at all" and 10 is "very sure". The 19 subscales are divided into three main categories, and the total score is the sum of these catagories. Higher value indicate better outcome. (Shaw et.al 2011).
Quality of Life (15D), health-related quality of life | Data collected during the interventions, baseline, 6 and 12 months.
  Mapping changes in 15D. The 15D is a generic, comprehensive (15-dimensional), self-administered instrument for measuring HRQoL. 5 ordinal levels on each dimension, by which more or less of the attribute is distinguished. A set of utility or preference weights is used to generate the 15D score (single index number) on a 0-1 scale. The valuation system of the 15D is based on an application of the multiattribute utility theory. The single index (15D score) on a 0 1 scale, representing the overall HRQoL (0 = being dead, 0.0162 = being unconscious or comatose, 1 = no problems on any dimension = 'full' HRQOL) is calculated from the health state descriptive system by using a set of population based preference or utility weights. (Harri Sintonen, http://www.15d-instrument.net).
Subjective somatic and psychological complaints | Data collected during the interventions, baseline, 6 and 12 months.
  Mapping changes with the scoring system subjective health complaints (SHC). The SHC consists of 29 questions concerning severity and duration of subjective somatic and psychological complaints. Intensity of each complaint is scored on a four-point scale from 0-3, where 0 is no complaints and three is severe complaints. The SHC inventory yields scores on single items and a total number of health complaints categorized into five factors: musculoskeletal pain (alpha=0.74), pseudoneurology (alpha=0.73), gastrointestinal problems (alpha=0.62), allergy (alpha=0.58) and flu (alpha=0.67). Eriksen HR, Ihlebæk C, Ursin H. A scoring system for subjective Health complaints (SHC). Scand J Public Health. 1999;27:63-72.
Vo2 peak | Data collected during the interventions, baseline and 12 months.
  Measured changes in the maximum amount of oxygen the participant can utilize during intense exercise. Measured in litres of oxygen per minute (L/min) or as a relative rate in (for example) millilitres of oxygen per kilogram of body mass per minute (e.g., mL/(kg·min). Physical test on a treadmill.
Body Mass Index | Data collected during the interventions, baseline, 6 and 12 months.
  Height will be added in Tanita MC-780U Multi Frequency Segmental Body Composition Analyzer. BMI will be reported in kg/m².
Waist circumstance (cm). | Data collected during the interventions, baseline, 6 and 12 months.
  Measured changes with Tanita MC-780U Multi Frequency Segmental Body Composition Analyzer.
Hight (centimetmeters) | Data collected during the interventions, baseline.
  The distance from the bottom of the feet to the top of the head, standing erect, measured with a stadiometer, in centimetres.
Promoting and hindering factors for Return to work. | Data collected during the interventions, baseline, 6 and 12 months.
  Mapping contextual conditions and mechanisms that might be important in the process back to work through In-Depth interviews

CONTACTS AND LOCATIONS:
Overall Officials: Geir Ove Vegsund, Study Director — Muritunet

IPD SHARING:
Plan to Share IPD: No
Abstract and lecture: Nordic Conference in Work and Rehabilitation. Abstract and lecture: Work Disability Prevention and Integration Conference 2019 An article in BMC Public Health, 2019, qualitative results. An article, mixed methods results, 2019